CLINICAL TRIAL: NCT04354129
Title: Safety, Tolerability, and Patient Satisfaction of 16.5% Subcutaneous Immunoglobulin (Cutaquig®) Treatment by Rapid Push in Patients With Primary or Secondary Immunodeficiency (PID or SID)
Brief Title: Observational Study of Subcutaneous Immunoglobulin (Cutaquig) in Patients With Primary and Secondary Immunodeficiency.
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00095620
Record Dates: First submitted 2020-04-08; First posted 2020-04-21 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Primary Immune Deficiency Disorder; Secondary Immune Deficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Immunoglobulins; Injections, Subcutaneous; Solutions; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At the infusion visits, blood samples will be collected for laboratory evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PID/SID Cutaquig Treated Patients: Immunoglobulin replacement therapy with subcutaneous injections of Cutaquig® 165 mg/mL at home.
  Interventions: Drug: Cutaquig®

INTERVENTIONS:
Drug: Cutaquig® — Immunoglobulin replacement therapy with subcutaneous injections of Cutaquig® 165 mg/mL at home.
  Other Names: Immunoglobulin (human) subcutaneous 16.5% Solution for injection (165 mg/mL)

SUMMARY:
This study will assess the relative safety, tolerability, and participant satisfaction in participants using the rapid manual push method with Cutaquig®. The hypothesis being that treatment with Cutaquig® by rapid manual push method will improve the safety, tolerability and patient satisfaction of participants with PID or SID.

Cutaquig® by rapid push is already approved in Canada and has proven to be efficacious in preventing significant infection. However, relative safety, tolerability, and patient satisfaction have not been studied in these patients. The information gained from this study will improve the safety and tolerability knowledge database and will support the optimal use of Cutaquig® - thus benefitting both physicians and patients.

DETAILED DESCRIPTION:
Primary and secondary immunodeficiency diseases (PID and SID, respectively) affect the development and/or function of the immune system, resulting in increased frequency of infection. Treatment of these disorders using Cutaquig® (a subcutaneous immunoglobulin infusion (SCIG)) was licensed in Canada in 2018 and has proven to be effective in preventing significant infection. Other brands of SCIG can be given by the participant using a syringe (called rapid manual push method), which shows the same efficacy as administration by a programmable pump. The rapid manual push method has the potential to improve quality of life, reduce infusion time, and reduce the cost of administration. This study will evaluate the safety, tolerability, and patient satisfaction of Cutaquig® by the rapid manual push method in participants with PID or SID. It will also compare the efficacy of Cutaquig with prior SCIG treatment, if applicable, in participants with PID or SID.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)
* Who have PID or SID requiring IgG replacement therapy
* For whom the investigator decides to maintain immunoglobulin replacement therapy with subcutaneous injections of Cutaquig® 165 mg/mL at home
* Having signed an informed consent form

Exclusion Criteria:

-Patients currently participating in another interventional study at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will observe approximately 30 adult patients with PID or SID requiring IgG replacement therapy, regardless of gender or treatment regimen. Patients will be enrolled from about 2-5 centres in Canada.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Safety of Infusion Rate | 6 months
  1. The primary objective is to assess safety of cutaquig® in patients with PID or SID by rapid push at infusion volumes ranging from 15 mL/infusion site to a maximum of 60 mL/infusion site into a maximum of 4 infusion sites and
  2. assess safety of a maximum infusion speed of 120 mL/h for all sites combined (2 mL/min)
Tolerability of Infusion Rate | 6 months
  1. The primary objective is to assess tolerability of cutaquig® in patients with PID or SID by rapid push at infusion volumes ranging from 15 mL/infusion site to a maximum of 60 mL/infusion site into a maximum of 4 infusion sites and
  2. assess tolerability of a maximum infusion speed of 120 mL/h for all sites combined (2 mL/min)

SECONDARY OUTCOMES:
Questionnaire | 6 months
  Key secondary objectives are to assess by a questionnaire
  1. time to infuse cutaquig®
  2. total volume infused per infusion site
  3. total volume infused per infusion
  4. frequency of infusion
  5. number of injection sites
  6. ease of infusion (injectability) Other secondary objectives are to
  7. assess patient quality of life (QoL) and patient satisfaction by using the EQ-5D-5L (descriptive system compromises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety and depression).
  8. compare the injectability of cutaquig® with prior SCIG administration if applicable

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Ritchie, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada